CLINICAL TRIAL: NCT02707185
Title: Physicians in Training and Critical Care Nurses Performance in Medical Code Events: Effect of Simulation-Based Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10-080; MCT STUDY (Other Grant/Funding Number: NEW YORK STATE ECRIP 2009)
Record Dates: First submitted 2011-05-10; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Ventricular Fibrillation
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physicians (Other): Physician in training:
  All internal medicine (IM), emergency medicine (EM), anesthesia (A), surgery (S) residents and all hospital ICU nurses.
  Interventions: Behavioral: Simulation-Based Training
- Nurses (Other): Nurses in Training
  Interventions: Behavioral: Simulation-Based Training

INTERVENTIONS:
Behavioral: Simulation-Based Training — An objective assessment tool has been developed and tested in medical code scenarios during training sessions recently done in the simulation lab. The tool has five domains: Airway, Breathing, Circulation, Communications/Leadership, and Defibrillation. Each domain consists of 3-8 tasks and skills.

SUMMARY:
METHODS:

Subjects:

All internal medicine (IM), emergency medicine (EM), anesthesia (A), surgery (S) residents and all hospital ICU nurses (approximately 400 subjects) will be undergoing evaluation and training in CPR techniques according to their department training policy.

Study Assessment Tool:

An objective assessment tool has been developed and tested in medical code scenarios during training sessions recently done in the simulation lab. The tool has five domains: Airway, Breathing, Circulation, Communications/Leadership, and Defibrillation. Each domain consists of 3-8 tasks and skills (attachment A).

Design:

* Phase I: In groups of five to six subjects, residents and nurses will undergo baseline assessment in CPR techniques in the simulation lab. Subject will be presented with a clinical scenario that includes cardiopulmonary arrest. Subjects will be scored by observers based on the previously described assessment tool and will be video recorded.
* Phase II: All study subjects who completed phase I assessment will undergo standardized debriefing and demonstration of proper CPR techniques after reviewing their individual baseline videotape followed by repeated demonstration in CPR techniques during a clinical scenario with cardiopulmonary arrest in the simulation lab. Knowledge retention will be assessed periodically.
* Phase III: Rates of survival to hospital discharge and survival at 24 hours in hospitalized patients after cardiopulmonary arrest collected by the CPR committee and QA department longitudinally for one year after completion of project training (phase II) will be reviewed and compared to the same period one year earlier (CPR outcome data are being collected since 2005 at St. Luke's-Roosevelt Hospitals).

ELIGIBILITY:
Inclusion Criteria:

* Physicians in training and nurses

Exclusion Criteria:

* Physicians in training and nurses refusing to have their data included in final analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Performance scale | Baseline and 1 year
  Change in performance scale at 1 year as compared to baseline
Rates of survival | 1 year
  Rates of survival to hospital discharge after cardiopulmonary arrest one year after completion of the simulation based training in CPR

SECONDARY OUTCOMES:
Survey questionnaire | Baseline and 1 year
  Change in survey questionnaire score at 1 year as compared to baseline. The questionnaire consists of 4 parts, including: adequacy of training, sense of preparedness, supervision and feedback, and general information. With the exception of the section on general information, responses are scored on a 5 point Likert scale.
Perceptions of preparedness | Baseline and 1 year
  Change in perceptions of preparedness at 1 year as compared to baseline. The method of assessment for this outcome measure is the Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Khouli, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's Roosevelt Roosevelt, New York, New York, United States